CLINICAL TRIAL: NCT01102907
Title: Beverages and Obesity: Effect of Food Form on Satiety and Hunger
Brief Title: Effect of Food Form on Satiety and Gastric Emptying
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1003M78873
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Appetite
Keywords: Appetite; Satiety; Gastric Emptying Time; Food Intake; Food Form

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Liquid Meal
  Interventions: Other: Liquid Breakfast
- Solid Meal
  Interventions: Other: Solid Breakfast Meal

INTERVENTIONS:
Other: Liquid Breakfast — The liquid breakfast meal will contain 370 calories and will consist of fruit juices and skim milk
  Groups: Liquid Meal
Other: Solid Breakfast Meal — The solid breakfast will contain 370 calories and will consist of oatmeal, golden delicious apples, blueberries, skim milk, and brown sugar.
  Groups: Solid Meal

SUMMARY:
Our objective is to determine whether food form (liquid vs. solid) alters gastric emptying, satiety, and food intake, when all macronutrients and fiber are controlled. The study population will include 10 healthy women, who have a normal body mass index. We have chosen to evaluate only women because this is a small pilot study and one of our endpoints is gastric emptying. Gastric emptying is known to differ between men and women. Gastric emptying will be evaluated using the Smartpill technology, satiety will be evaluated using computerized visual analog scales/questions, and food intake will be measured by providing subjects with an ad libitum/buffet-style lunch.

Our hypothesis is that our subjects will be less hungry after they eat a solid breakfast compared to a liquid breakfast. We also hypothesize that our subjects will have a slower gastric emptying time after they eat the solid meal. Lastly, we think subjects will want to eat less food at lunch time if they have eaten a solid meal compared to a liquid meal for breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* Age 18 - 35
* Body mass index in the healthy range between 18.5 and 25
* Proficient English speakers
* Non-smoking
* Not taking medications
* Non-dieting (weight stable over last 3 months)
* Able to swallow a large capsule

Exclusion Criteria:

* Irregular or erratic breakfast eating patterns
* Food allergies to ingredients commonly found in test products or pizza
* Distaste for test products or pizza
* BMI less than 18.5 or greater than 25
* Weight change > 5 kg in last 3 months (intentional or unintentional)
* Difficulty swallowing
* Cardiovascular disease
* Diabetes mellitus (fasting blood sugar > 126 mg/dl)
* Cancer in prior 5 years (except basal cell carcinoma of skin)
* Kidney or liver disease
* Any gastrointestinal conditions that may affect digestion and absorption
* Recent bacterial infection (< 3 months)
* Chronic medication use
* History of drug or alcohol abuse in prior 6 months
* Concurrent or recent intervention study participation
* Vegetarians or people who ate more than approximately 15 g of fiber per day
* Pregnant or lactating women
* Women with irregular menstrual cycles

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women; age 18 - 35; body mass index in the healthy range between 18.5 and 25; proficient English speakers; non-smoking; not taking medications; non-dieting (weight stable over last 3 months); able to swallow a large capsule
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Determine whether food form (liquid vs. solid) alters gastric emptying time when all macronutrients and fiber are controlled. | May 2010 to December 2010
  Subjects will consume both liquid and solid meals and we will evaluate and compare gastric emptying time after each of them.

SECONDARY OUTCOMES:
Determine whether food form (liquid vs. solid) alters satiety and food intake when all macronutrients and fiber are controlled. | May 2010 to December 2010
  Subjects will consume both liquid and solid meals and we will evaluate and compare appetite and food intake after each of them.

CONTACTS AND LOCATIONS:
Overall Officials: Holly J Willis, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Saint Paul, Minnesota, United States